CLINICAL TRIAL: NCT01896011
Title: Effect of Teriparatide on Fracture Healing in Patients With Incomplete Atypical Femur Fractures: a Randomized Controlled Trial
Brief Title: Effect of Teriparatide on Fracture Healing in Patients With Incomplete Atypical Femur Fractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-0170; Control # 164050 (Registry Identifier: Health Canada BGTD)
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Non Displaced Atypical Femoral Fractures
MeSH Terms: interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriparatide 20 mcg daily (Active Comparator): Teriparatide (Forteo) 20 mcg daily by injection pen for 12-24 months
  Interventions: Biological: Teriparatide 20 mcg
- Placebo (Placebo Comparator): Placebo injection pen identical to active drug injection pen
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Teriparatide 20 mcg — Teriparatide 20 mcg injection pen
  Other Names: Brand name Forteo
  Arms: Teriparatide 20 mcg daily
Other: Placebo — Placebo 20 mcg injection pen
  Arms: Placebo

SUMMARY:
Atypical femur (thigh bone) fractures (AFFs) are uncommon low-trauma fractures which often occur without warning, are highly debilitating, and are slow to heal. As physicians learn more about them, AFFs are increasingly being identified prior to a total break. However, there's no evidence on the best way to treat these non-displaced AFFs. One option is teriparatide, an osteoporosis medication that can build new bone. Investigators will conduct a double blind randomized placebo controlled trial to examine whether teriparatide use in AFF patients with an incomplete break will help accelerate fracture healing and prevent surgical intervention. Co-primary outcomes include change in WOMAC scores from baseline to 12 months and number of participants requiring surgical intervention at 12 months. Investigators will recruit 60 women and men over the age of 30 who have experienced an incomplete AFF. Participants will be randomly assigned to either teriparatide (20 mcg/day) or placebo (using an identical injection pen) for up to 2 years. As AFFs are highly debilitating, a trial examining the use of Teriparatide in this population is urgently needed.

ELIGIBILITY:
Inclusion Criteria:

i. Female or male; ii. Over the age of 30; iii. Experienced an incomplete AFF that satisfies the diagnostic criteria as set forth by the American Society for Bone and Mineral Research (ASBMR) International Task Force on AFFs:

1. Atraumatic or low trauma incomplete stress fractures, defined as fractures sustained with minimal force, such as a fall from standing height;
2. From distal to the lesser trochanter to proximal to the supracondylar flare along the femoral shaft.
3. Radiographic confirmation of AFF features is required for a definitive diagnosis. Incomplete AFF features include cortical thickening, cortical beaking, and lucency line. Patients with cortical beaking without lucency line can be included.

Exclusion Criteria:

i. Peri-prosthetic fractures, ii. High trauma fractures, iii. Pathological fractures secondary to metastases or metabolic bone diseases other than osteoporosis, iv. Fractures that are not confirmed by radiological investigations, v. Contraindication to use of teriparatide such as:

1. pregnant or nursing mothers, or women who are planning on pregnancy within 1 year of completing teriparatide therapy,
2. hypersensitivity to teriparatide,
3. severe renal impairment,
4. multiple myeloma,
5. active cancer in past 5 years (other than non-melanoma skin cancer),
6. primary hyperparathyroidism,
7. hypercalcemia,
8. Paget's disease or other conditions that may increase the risk for osteosarcoma,
9. Prior radiation therapy involving the skeleton, vi. Concomitant use of other osteoporosis therapies including bisphosphonates or denosumab (except calcitonin).

AFF patients with complete fractures on the contralateral side or patients with secondary osteoporosis will not be excluded.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in the modified The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)of the affected limb (the femur that has the incomplete AFF) | baseline to 12 months
The proportion of patients requiring surgical intervention | baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD, PhD, Study Director — University Health Network, Toronto; Lianne E Tile, Md, MEd, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada